CLINICAL TRIAL: NCT06058039
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Oral NMRA-335140 Versus Placebo in Participants With Major Depressive Disorder
Brief Title: Study to Assess the Effects of Oral NMRA-335140 in Participants With Major Depressive Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neumora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRA-335140-303; KOASTAL-3 (Other: Neumora Therapeutics)
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; NMRA-335140; Placebo-controlled; Double-blind; Navacaprant; NMRA335140; NMRA 335140
MeSH Terms: conditions — Depressive Disorder, Major | interventions — BTRX-335140

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor will also be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NMRA-335140 80 milligrams (mg) once daily (QD) (Experimental): Participants will receive a NMRA-335140 tablet at a dose of 80 mg QD
  Interventions: Drug: NMRA-335140
- Placebo (Placebo Comparator): Placebo participants will receive matching placebo tablet once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NMRA-335140 — Participants will receive NMRA-335140 at a dose of 80 mg QD, orally
  Other Names: BTRX-335140; CYM-53093; Navacaprant
  Arms: NMRA-335140 80 milligrams (mg) once daily (QD)
Drug: Placebo — Placebo will be administered orally
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, multicenter study will evaluate the effects of NMRA-335140 (formerly BTRX-335140) on symptoms of depression in participants with Major Depressive Disorder (MDD). The study design consists of a Screening Period (up to 35 days), and a 6-week Treatment Period (during which participants will receive either NMRA-335140 or placebo). At the completion of the 6-week Treatment Period, participants who complete the study, provide informed consent, and meet the eligibility criteria may enter an open-label extension study (NMRA-335140-501).

ELIGIBILITY:
Key Inclusion Criteria:

* Have a primary Diagnostic and Statistical Manual of Mental Disorders Fifth Edition Text Revised (DSM-5-TR) diagnosis of MDD without psychotic features confirmed by Structured Clinical Interview for DSM 5 Disorders, Clinical Trials Version (SCID 5 CT) at screening (this may be a first or recurrent episode).
* Participant's current major depressive episode must be confirmed by independent assessment.
* The symptoms of the current MDD episode have been present for more than 4 weeks prior to the Screening Visit, but no longer than 12 months prior to the Screening Visit.
* Have a MADRS total score of 25 or higher at Screening and Baseline.
* A change in MADRS total score between Screening and Baseline of ≤20%.

Key Exclusion Criteria:

* Have failed 2 or more courses of antidepressant treatment at sufficient doses for at least 6 to 8 weeks for the current MDD episode.
* Currently or in the past year have been diagnosed with a personality disorder per the DSM-5-TR or in the past 3 years have been diagnosed with any of the following DSM-5-TR disorders: anorexia nervosa, bulimia nervosa, or binge eating disorder. Participants with comorbid generalized anxiety disorder, social anxiety disorder, simple phobias, or panic disorder for whom MDD is considered the primary diagnosis are not excluded.
* Have a lifetime diagnosis of bipolar 1 or 2, schizophrenia, schizoaffective, schizophreniform, obsessive compulsive disorder, or post-traumatic stress disorder (PTSD).
* Have moderate to severe substance or alcohol use disorder, per DSM-5-TR criteria, within the 12 months prior to screening (excluding nicotine).
* Are actively suicidal (eg, any suicide attempts within the past 12 months) or are at serious suicidal risk as indicated by any current suicidal intent, including a plan, as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) (score of "YES" on suicidal ideations Item 4 or 5 within 3 months prior to Visit 1 [Screening]) and/or based on clinical evaluation by the Investigator; or are homicidal, in the opinion of the Investigator. Participants who are currently hospitalized for MDD symptoms or suicidality are not allowed into the study. If there is a recent history (within 3 months of screening) of hospitalization due to MDD symptoms, the participant should be discussed with the Medical Monitor for eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 6 in the Montgomery-Asberg Depression Rating Scale (MADRS) total score | Baseline and up to Week 6
  The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants are rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item will be scored on a 7- point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity. Thus, scores in the MADRS range from 0 to 60, with increasing scores indicating increasing severity.

SECONDARY OUTCOMES:
Change from Baseline to Week 6 assessed in the Snaith-Hamilton Pleasure Scale (SHAPS) total score | Baseline and up to Week 6
  The SHAPS is a 14-item participant-reported instrument which measures anhedonia. It has been shown to be valid and reliable in normal and clinical samples, with adequate construct validity, satisfactory test-retest reliability, and high internal consistency. The scale will be completed by the participant and reviewed by site personnel qualified to oversee completeness. Each of the 14 items has a set of 4 responses, 2 of which endorse agreement (Definitely Agree, Agree) and 2 of which endorse disagreement (Disagree, Strongly Disagree). A total score can be derived by summing the response items; where those answered with "strongly agree" will be coded as a 1, while a "strongly disagree" response will be coded as 4. Therefore, scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.

CONTACTS AND LOCATIONS:
Locations (63):
- United States (31):
  - Neumora Investigator Site, Cerritos, California
  - Neumora Investigator Site, Irvine, California
  - Neumora Investigator Site, Long Beach, California
  - Neumora Investigator Site, San Diego, California
  - Neumora Investigator Site, San Francisco, California
  - Neumora Investigator Site, New Haven, Connecticut
  - Neumora Investigator Site, Brandon, Florida
  - Neumora Investigator Site, Hialeah, Florida
  - Neumora Investigator Site, Jacksonville, Florida
  - Neumora Investigator Site, Miami, Florida
  - Neumora Investigator site, Miami, Florida
  - Neumora Investigator Site, Miami Beach, Florida
  - Neumora Investigator site, Miami Springs, Florida
  - Neumora Investigator Site, Palm Bay, Florida
  - Neumora Investigator Site, Pembroke Pines, Florida
  - Neumora Investigator Site, Pompano Beach, Florida
  - Neumora Investigator Site, Saint Augustine, Florida
  - Neumora Investigator Site, Atlanta, Georgia
  - Neumora Investigator Site, Decatur, Georgia
  - Neumora Investigator Site, Savannah, Georgia
  - Neumora Investigator Site, Springfield, Massachusetts
  - Neumora Investigator Site, St Louis, Missouri
  - Neumora Investigator Site, Omaha, Nebraska
  - Neumora Investigator Site, Berlin, New Jersey
  - Neumora Investigator Site, New York, New York
  - Neumora Investigator Site, Staten Island, New York
  - Neumora Investigator Site, Charlotte, North Carolina
  - Neumora Investigator Site, Austin, Texas
  - Neumora Investigator Site, DeSoto, Texas
  - Neumora Investigator Site, Fort Worth, Texas
  - Neumora Investigator Site, Plano, Texas
- Bulgaria (7):
  - Neumora Investigator Site, Cherven Bryag, Pleven
  - Neumora Investigator Site, Sofia, Sofia-Grad
  - Neumora Investigator Site, Kardzhali
  - Neumora Investigator Site, Pleven
  - Neumora Investigator Site, Targovishte
  - Neumora Investigator Site #1, Varna
  - Neumora Investigator Site, Varna
- Czechia (5):
  - Neumora Investigator Site, Pilsen, Plzen
  - Neumora Investigator Site, Prague, Prague
  - Neumora Investigator Site #1, Kladno, South Bohemian
  - Neumora Investigator Site, Kladno
  - Neumora Investigator Site, Prague
- Finland (3):
  - Neumora Investigator Site, Helsinki, Etelä-Suomen Lääni
  - Neumora Investigator Site, Turku, Etelä-Suomen Lääni
  - Neumora Investigator Site, Oulu, Oulun Lääni
- France (6):
  - Neumora Investigator Site, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Neumora Investigator Site, Douai, Hauts-de-France
  - Neumora Investigator Site, Montpellier, Hérault
  - Neumora Investigator Site, Angers, Maine-et-Loire
  - Neumora Investigator Site, La Roche-sur-Yon, Vendée
  - Neumora Investigator Site, Poitiers, Vienne
- Germany (3):
  - Neumora Investigator Site #1, Berlin
  - Neumora Investigator Site, Berlin
  - Neumora Investigator Site, Hamburg
- Poland (6):
  - Neumora Investigator Site, Suchy Las, Greater Poland Voivodeship
  - Neumora Investigator Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Neumora Investigator Site, Wroclaw, Lower Silesian Voivodeship
  - Neumora Investigator Site, Lublin, Lublin Voivodeship
  - Neumora Investigator Site, Bialystok, Podlaskie Voivodeship
  - Neumora Investigator Site, Gdansk, Pomeranian Voivodeship
- Sweden (2):
  - Neumora Investigator Site, Lund, Skåne County
  - Neumora Investigator Site, Stockholm, Stockholm County

IPD SHARING:
Plan to Share IPD: No